CLINICAL TRIAL: NCT06456541
Title: Determination of Hypoallergenicity of an Extensively Hydrolyzed Infant Formula in Infants and Children With Cow's Milk Allergy
Brief Title: Infant Formula in Infants and Children With Cow's Milk Allergy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AL60
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Extensively Hydrolyzed Formula (Experimental): Administered during food challenge and at home feeding period of 7 days
  Interventions: Other: Experimental Extensively Hydrolyzed Formula
- Placebo Extensively Hydrolyzed Formula (Placebo Comparator): Administered during food challenge
  Interventions: Other: Placebo Extensively Hydrolyzed Formula

INTERVENTIONS:
Other: Experimental Extensively Hydrolyzed Formula — Experimental powder formula
  Arms: Experimental Extensively Hydrolyzed Formula
Other: Placebo Extensively Hydrolyzed Formula — Placebo powder formula
  Arms: Placebo Extensively Hydrolyzed Formula

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled food challenge to be conducted in infants and children with confirmed IgE-mediated cow's milk allergy (CMA), followed by a 7-day open feeding of the experimental formula.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s) is/are willing for their child to undergo confirmatory testing or must have had at least one of the following within 6 months of enrollment:

  1. Physician diagnosis of IgE-mediated CMA, according to the participant's clinical history (e.g. gastrointestinal symptoms, hives, respiratory symptoms or angioedema) AND, detectable serum milk-specific IgE >0.7 kUᴀ/L or positive skin prick test wheal ≥5 mm;
  2. Documentation of milk-specific serum IgE >15 kUᴀ/L or > 5 kUᴀ/L if younger than 1 year;
  3. Documented cow's milk skin prick test wheal >10mm;
  4. Physician-supervised oral food challenge that elicited immediate, objective, allergic symptoms.
* Participant's parent(s) agree for their child to stop oral steroid use within 14 days and antihistamine use within 7 days prior to confirmation of diagnosis and food challenges.
* Participant had followed a strict cow's milk protein-free diet for at least 2 weeks prior to enrollment.
* Parent(s) confirm their intention not to administer any products containing cow's milk protein during the study.
* Participant is between 3 months and 12 years of age at enrollment.
* Participant's parent(s) has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* Participant is partially or exclusively breastfed at the time of enrollment.
* Participant is consuming an amino acid-based formula due to failure on an extensively hydrolyzed formula.
* Significant chronic medical diseases including major chromosomal or congenital anomalies, gastrointestinal diseases, or abnormalities other than CMA, immunodeficiencies, unstable asthma, eczema and/or food allergies treated with biologics (omalizumab or other monoclonal antibody), FPIES, eosinophilic esophagitis, and severe uncontrolled eczema.
* Previous severe anaphylactic reaction to cow's milk within the last two years.,
* An adverse medical history or current condition that is thought by the investigator to have potential for effects on tolerance or the hypoallergenicity test.
* Participant has an allergy or intolerance to any ingredient in the study product, as reported by the parent.
* Participant is consuming baked milk products.
* Use of and/or changing dose of high potency steroids.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Food Challenge Reactions | Food Challenge 1 to Food Challenge 2 (within 14 days of the Food Challenge 1) (followed by 7 days of feeding the experimental formula at home.)
  Percent of positive food challenge reactions to the experimental formula administered to cow's milk allergic infants and children.

SECONDARY OUTCOMES:
Volume of Experimental Formula Intake | Home Feeding Day 1 to Day 7
  Parent completed diaries of Intake
Food Intake during Study | Home Feeding Day 1 to Day 7
  Parent completed daily food diaries
Gastrointestinal Symptoms | Home Feeding Day 1 to Day 7
  Parent completed diaries
Medication Use | Home Feeding Day 1 to Day 7
  Parent completed diaries
Food Challenge Positive Reactions | Home Feeding Day 1 to Day 7
  Percent of positive food challenge reactions to the experimental formula

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Michigan Food Allergy Clinic, Ann Arbor, Michigan
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No